CLINICAL TRIAL: NCT02876484
Title: Effects of Chenodeoxycholic Acid and Colesevelam on GLP-1 Secretion, During a Meal, After Roux-en-Y Gastric Bypass
Brief Title: Effects of Bile Acids and Bile Acid Sequestrants on GLP-1 Secretion After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Saur Svane, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IJ-G2-16
Record Dates: First submitted 2016-07-01; First posted 2016-08-23 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Colesevelam Hydrochloride; Chenodeoxycholic Acid; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Experimental): Morning meal: brown bread, margarine, cheese, yoghurt, oatmeal, raisins, almonds, water, PCM.
  25 ml water
  Interventions: Other: Water
- Chenodeoxycholic Acid (Experimental): Morning meal: brown bread, margarine, cheese, yoghurt, oatmeal, raisins, almonds, water, PCM. Chenodeoxycholic acid (1250 mg) mixed in 25 ml yoghurt
  Interventions: Drug: Chenodeoxycholic Acid
- Colesevelam (Experimental): Morning meal: brown bread, margarine, cheese, yoghurt, oatmeal, raisins, almonds, water, PCM. Colesevelam (3,75 g) dissolved in 25 ml water and mixed in 25 ml yoghurt.
  Interventions: Drug: Colesevelam
- Colesevelam x 2 (Experimental): plus (on another study day) 3,75 g colesevelam administered the evening before the experiment. Morning meal: brown bread, margarine, cheese, yoghurt, oatmeal, raisins, almonds, water, PCM. Colesevelam (3,75 g) dissolved in 25 ml water and mixed in 25 ml yoghurt.
  Interventions: Drug: Colesevelam

INTERVENTIONS:
Drug: Colesevelam
  Arms: Colesevelam; Colesevelam x 2
Drug: Chenodeoxycholic Acid
  Arms: Chenodeoxycholic Acid
Other: Water
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of bile acid and bile acids sequestrants on GLP-1 Secretion, during a meal, in patients after Roux-en-Y gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated RYGB performed minimum 3 months prior to the study.
* Fasting plasma glucose < 7,0 mM, HbA1c < 48 mmol/mol 3 months after RYGB

Exclusion Criteria:

* Fasting plasma glucose > 7,0 mM, HbA1c > 48 mmol/mol 3 months after RYGB.
* Dysregulated thyroid diseases, use of antithyroid treatment.
* Late diabetic complications as retinopathy, renal insufficiency, neuropathy or previous pancreatitis.
* Complications to RYGB. Documented reactive hypoglycaemia, severe dumping (vomiting, diarrhea, severe abdominal pain after food intake).
* Cholecystectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
GLP-1 secretion (evaluated by iAUC) | -10, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes after mixed meal

SECONDARY OUTCOMES:
Glucose levels | -10, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
Insulin secretion | -10, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
PYY secretion | -10, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
Bile acids/FGF19 concentrations | -10, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
Appetite measurements (VAS-score) | 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
PCM levels | Baseline, 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240 minutes
C-peptide secretion | Baseline, 0, 5, 10, 20, 30, 45, 60, 90, 120, 180, 240 minutes
Glucagon secretion | Baseline, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 minutes
GIP secretion | 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
CCK secretion | 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
Ghrelin | 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes
Total bile acid secretion | 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes